CLINICAL TRIAL: NCT04221204
Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetics Profiles and Preliminary Efficacy of 3D185 Monotherapy in Subjects With Advanced Solid Tumors
Brief Title: A Monotherapy in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 3D Medicines (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3D185-CN-001
Record Dates: First submitted 2019-12-13; First posted 2020-01-09 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Intervention Model Description: sequential assignment The starting dose in this dose-escalation study is 50 mg, and the preset 6 dose-escalation cohorts are 50 mg, 100 mg, 150 mg, 200 mg, 250 mg, and 300 mg, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label, Dose-Escalation (Experimental): The starting dose in this dose-escalation study is 50 mg, and the preset 6 dose-escalation cohorts are 50 mg, 100 mg, 150 mg, 200 mg, 250 mg, and 300 mg, respectively. This study adopts an i3+3 method for dose escalation.
  All subjects in each cohort will receive a single oral dose of 3D185, followed by a 7-day washout period (i.e. single-dose PK study period). Then, subjects will receive consecutive daily doses (Once daily [QD], 28 days/cycle) until disease progression, death, unacceptable toxicity, or withdraw of informed consent, whichever comes first
  Interventions: Drug: Highly selective FGFR1-3 inhibitor

INTERVENTIONS:
Drug: Highly selective FGFR1-3 inhibitor — All subjects in each cohort will receive a single oral dose of 3D185, followed by a 7-day washout period (i.e. single-dose PK study period). Then, subjects will receive consecutive daily doses (Once daily [QD], 28 days/cycle) until disease progression, death, unacceptable toxicity, or withdraw of informed consent, whichever comes first. The dose limiting toxicity (DLT) evaluation period includes the single-dose PK study period and the first treatment cycle (within 35 days after the first dose). The enrolled subjects will be sequentially assigned to the planned dose cohorts according to the protocol and receive 3D185 treatment to observe the occurrence of DLT.

SUMMARY:
A Phase 1 Study of the Safety, Tolerability, Pharmacokinetics Profiles, and Preliminary Efficacy of 3D185 Monotherapy in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
Subjects with advanced solid tumors who have no available standard therapy or who have failed standard therapies.

This is an open-label, global multicenter, dose-escalation phase 1 study of safety, tolerability, preliminary PK profile, and preliminary efficacy of 3D185 capsules monotherapy in subjects with advanced solid tumors.

The starting dose in this dose-escalation study is 50 mg, and the preset 6 dose-escalation cohorts are 50 mg, 100 mg, 150 mg, 200 mg, 250 mg, and 300 mg, respectively.

ELIGIBILITY:
Study Population:

In the study, male or female adult subjects ≥ 18 years of age, with advanced solid tumors with no prior standard therapy or failed to establish standard therapies are eligible.

Inclusion Criteria:

1. Subjects must be male or female and ≥ 18 years of age on the day of enrollment.
2. Subjects must have a histological diagnosis of locally advanced or metastatic malignant solid tumors. Subjects must have failed or have been intolerant to established standard therapies, or standard therapies did not exist or were no longer effective for a given tumor type, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds.
3. Subjects must have at least one evaluable lesion (according to RECIST 1.1, see Appendix 1);
4. ECOG Performance Status of 0 or 1.
5. Life expectancy ≥ 12 weeks.
6. Subjects must have normal levels of total serum calcium and total phosphate.
7. Subjects must have adequate organ and bone marrow function (no hematopoietic growth factor, blood transfusion, or platelet therapy within 1 week before the first dose):

   * CBC: neutrophils ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 9.0 g/dL.
   * Liver function: total bilirubin ≤ 1.5 × ULN; ALT/AST ≤ 2.5 × ULN without liver metastasis; ALT/AST ≤ 5 × ULN with liver metastasis;
   * Coagulation: International normalized ratio (INR) ≤ 1.5 × ULN and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (for patients undergoing anticoagulant therapy. The Investigator will judge that the INR and APTT are within a safe and effective treatment range).
   * Renal function: serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min/1.73 m2 in the condition of creatinine level > ULN; urine protein qualitative ≤ 1 + (if ≥ 2+, 24 hours of urine protein test is required, if 24 hours urine protein <1 g, then allowed to enroll);
   * Adequate cardiac function left ventricular ejection fraction (LVEF) > 50% for 2 dimensional cardiac ultrasound;
8. Subjects must have signed and dated an IRB/IEC approved written informed consent form that under regulatory and institutional guidelines, and this must be obtained before the performance of any protocol-related procedures.

Exclusion Criteria:

Subjects who meet any of the following criteria should be excluded from the study:

1. Subjects who received other investigational products or devices in other clinical trials within 4 weeks before the first dose;
2. Subjects who received anti-tumor therapy (except for mitomycin, nitrosourea, and fluorouracil oral drugs) within 4 weeks before the first dose, including but not limited to chemotherapy, radiotherapy (palliative radiotherapy is completed at least 2 weeks before the first dose can enroll), targeted therapy or immunotherapy.

   Note: Mitomycin and nitrosourea have been treated within 6 weeks after the last dose; oral fluorouracil such as tegafur and capecitabine has been treated within 2 weeks after the last dose.
3. Subjects who previously received FGFR1-3 specific inhibitor therapy.
4. Subjects who have previous toxicity of anti-tumor therapy that has not been returned to level 0 or 1. (Alopecia, chemotherapy-induced peripheral neurotoxicity and ototoxicity ≤ Grade 2 can enroll);
5. Subjects who received a CYP3A4 and/or CYP2C8 strong inhibitor or a CYP3A4 strong inducer (see Appendix 6) within 7 days prior to the first dose, and need to continue using these drugs;
6. Subjects who have any of the following eye diseases/conditions:

   * History of retinal pigment epithelial detachment (RPED);
   * History of laser treatment or intraocular injection for macular degeneration;
   * History of dry or wet age-related macular degeneration;
   * History of retinal vein occlusion (RVO);
   * History of retinal degenerative diseases;
   * History of chorioretinal lesions;
7. Subjects who received clinical intervention for biliary obstruction 14 days prior to the first dose or the Investigator judges that the symptoms had not resolved or required anti-infective treatment.
8. Subjects who have gastrointestinal disorders that will affect oral administration or the Investigator judges that the absorption of 3D185 will be interfered.
9. Subjects underwent major surgery (except biopsy), or the surgical incision has not completely healed within 4 weeks prior to the first dose.
10. Subjects who had clinically uncontrollable pleural effusion, ascites, or pericardial effusion within 2 weeks prior to the first dose.
11. Subjects who have symptomatic brain metastases or spinal cord compression. Subjects who have previously treatment for brain metastases, if the clinical condition is stable and imaging evidence does not show disease progression within 4 weeks prior to the first dose, and do not need corticosteroid treatment within 2 weeks prior to the first dose, can enroll.
12. Subjects who have active bacterial or fungal infections (CTCAE ≥ 2) that required systemic treatment within 14 days prior to the first dose.
13. Subjects who have active HBV infection (Tests should include assessment of HBsAg and HBc IgG antibody. If one parameter is positive, determine HBV-DNA to confirm acute infection. Patients with positive results for HBsAg and/or HBV-DNA are considered active HBV infection) and/or active HCV infection (HCV antibody testing positive);
14. Subjects who have clinically significant cardiovascular diseases that occurred 6 months prior to enrollment. Cardiovascular diseases include, but not limited to follows:

    * Acute myocardial infarction;
    * Severe/unstable angina;
    * Cerebrovascular accident or transient ischemic attack;
    * Congestive heart failure (New York Heart Association > Class II, see Appendix 3);
    * Arrhythmias that require antiarrhythmic treatment except for beta blockers or digoxin;
    * Repeated ECG with QTc interval > 450 ms;
    * High blood pressure that cannot be controlled by antihypertensive drugs (systolic blood pressure > 150 mm Hg, diastolic blood pressure > 100 mmHg).
15. Subjects who have clinically significant abnormal serum electrolytes (Patients must have corrected calcium and phosphate < institutional ULN).
16. Subjects who are receiving warfarin (low-dose warfarin as 2 mg/day is acceptable); or receiving antiplatelet anticoagulant therapy (aspirin at dose ≥300 mg/day, clopidogrel at dose ≥75 mg/day).
17. Female subjects in pregnancy or lactation. Male subjects or female subjects at reproductive ages who are unwilling to receive effective contraceptive measures.
18. Subjects who are judged by the Investigator to be unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation: frequency and severity of AEs | 24 months
  Evaluated based on the frequency and severity of AEs according to NCI CTCAE v4.03.
Tolerability Evaluation: frequency and severity of AEs | 24 Months
  based on the frequency and severity of AEs according to NCI CTCAE v4.03.

SECONDARY OUTCOMES:
Efficacy evaluation: Complete Response | 24 months
  Per RECIST version 1.1 criteria in Solid tumors v 1.1 (RECIST) assessed by investigator
Pharmacokinetics (PK) evaluation: Cmax (mg/L) | 24 months
  The test of PK samples will be performed by central laboratory. The PK parameters will be calculated using standard non-compartment models and WinNonlin® Professional 6.4 or higher version (Certara, Princeton, NJ, USA) or SAS® 9.3 or higher version (SAS Institute, Inc., Cary, North Carolina) to fully reflect the drug absorption, distribution and elimination characteristics in the human body. The interim PK parameters will be calculated using the planned blood collection time, and the final PK parameters will be calculated using the actual blood collection time.
PK evaluation: Tmax (minutes) | 24 months
  The test of PK samples will be performed by central laboratory. The PK parameters will be calculated using standard non-compartment models and WinNonlin® Professional 6.4 or higher version (Certara, Princeton, NJ, USA) or SAS® 9.3 or higher version (SAS Institute, Inc., Cary, North Carolina) to fully reflect the drug absorption, distribution and elimination characteristics in the human body. The interim PK parameters will be calculated using the planned blood collection time, and the final PK parameters will be calculated using the actual blood collection time.
PK evaluation: AUC0-24 h, AUC0-96 h, AUC0-∞, | 24 months
  The PK parameters will be calculated using standard non-compartment models and WinNonlin® Professional 6.4 or higher version (Certara, Princeton, NJ, USA) or SAS® 9.3 or higher version (SAS Institute, Inc., Cary, North Carolina) to fully reflect the drug absorption, distribution and elimination characteristics in the human body. The interim PK parameters will be calculated using the planned blood collection time, and the final PK parameters will be calculated using the actual blood collection time.
PK evaluation: t1/2 | 24 months
  The test of PK samples will be performed by central laboratory. The PK parameters will be calculated using standard non-compartment models and WinNonlin® Professional 6.4 or higher version (Certara, Princeton, NJ, USA) or SAS® 9.3 or higher version (SAS Institute, Inc., Cary, North Carolina) to fully reflect the drug absorption, distribution and elimination characteristics in the human body. The interim PK parameters will be calculated using the planned blood collection time, and the final PK parameters will be calculated using the actual blood collection time.
PK evaluation: Clearance | 24 months
  The test of PK samples will be performed by central laboratory. The PK parameters will be calculated using standard non-compartment models and WinNonlin® Professional 6.4 or higher version (Certara, Princeton, NJ, USA) or SAS®9.3 or higher version (SAS Institute, Inc., Cary, North Carolina) to fully reflect the drug absorption, distribution and elimination characteristics in the human body. The interim PK parameters will be calculated using the planned blood collection time, and the final PK parameters will be calculated using the actual blood collection time.
PK evaluation: Vd. | 24 months
  The test of PK samples will be performed by central laboratory. The PK parameters will be calculated using standard non-compartment models and WinNonlin® Professional 6.4 or higher version (Certara, Princeton, NJ, USA) or SAS® 9.3 or higher version (SAS Institute, Inc., Cary, North Carolina) to fully reflect the drug absorption, distribution and elimination characteristics in the human body. The interim PK parameters will be calculated using the planned blood collection time, and the final PK parameters will be calculated using the actual blood collection time.
Progressive Disease evaluation | 24 months
  assessed by analyzing the change in serum phosphate levels relative to baseline level over time (Serum biochemistry test).
Efficacy evaluation: Partial Response | 24 months
  Per RECIST version 1.1 criteria in Solid tumors v 1.1 (RECIST) assessed by investigator
Efficacy evaluation: Stable Disease | 24 months
  Per RECIST version 1.1 criteria in Solid tumors v 1.1 (RECIST) assessed by investigator
Efficacy evaluation: Disease Progression | 24 months
  assessed by analyzing the change in serum phosphate levels relative to baseline level over time (Serum biochemistry test).
Objective Response Rale (ORR) (CR+PR) | 24 months
  Per RECIST version 1.1 criteria in Solid tumors v 1.1 (RECIST) assessed by investigator
disease control rate (DCR) (CR+PR+SD) | 24 months
  Per RECIST version 1.1 criteria Per RECIST version 1.1 criteria in Solid tumors v 1.1 (RECIST) assessed by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Di Zhu, Study Director — 3D Medicines (Beijing) Co., Ltd.
Locations (2):
- Sarcoma Oncolog Research Center, Santa Monica, California, United States
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No